CLINICAL TRIAL: NCT00498212
Title: A Phase 2, Single-Blind, Randomized Study of Safety and Immunogenicity Following Vaccination With Single or Double Doses of HEPLISAV™ in Adults With End-Stage Renal Disease
Brief Title: A Safety and Efficacy Study of a Single or Double Dose of HEPLISAV™ Hepatitis B Vaccine in Adults With End-Stage Renal Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Voluntary halt due to an FDA Clinical Hold issued in relation to DV2-HBV-10.
Sponsor: Dynavax Technologies Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DV2-HBV-11
Record Dates: First submitted 2007-07-05; First posted 2007-07-09 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Hepatitis B
Keywords: Heplisav; Hepatitis B; Hepatitis; HBV; Hepatitis B vaccine; kidney disease; renal disease; kidney failure; renal failure
MeSH Terms: conditions — Hepatitis B; Hepatitis; Kidney Diseases; Renal Insufficiency | interventions — Hepatitis B Vaccines

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1018 ISS-HBsAg-Single (Experimental): Single dose (3000 µg 1018 ISS + 20 µg rHBsAg)
  Interventions: Biological: 1018 ISS-HBsAg-Single
- 1018 ISS-HBsAg-Double (Experimental): Double dose (6000 µg 1018 ISS + 40 µg rHBsAg)
  Interventions: Biological: 1018 ISS-HBsAg-Double

INTERVENTIONS:
Biological: 1018 ISS-HBsAg-Single — Intramuscular (IM) injection at Day 0, Week 4 and Week 24
  Other Names: HEPLISAV™
  Arms: 1018 ISS-HBsAg-Single
Biological: 1018 ISS-HBsAg-Double — Intramuscular (IM) injection at Day 0, Week 4 and Week 24
  Other Names: HEPLISAV™
  Arms: 1018 ISS-HBsAg-Double

SUMMARY:
The purpose of this study is to find out if a new investigational hepatitis B virus (HBV) vaccine, HEPLISAV™, is safe and effective for end-stage renal disease (ESRD) patients. Two dose levels will be studied: a single dose and a double dose. We expect both dose levels to safely immunize patients against HBV. The study will determine which dose does this best.

DETAILED DESCRIPTION:
Infection with hepatitis B virus (HBV) is a major global health problem. Worldwide, it is estimated that 2 billion people have been infected previously and 350 million are chronically infected. While acute HBV infection is associated with significant illness, the risk of chronic infection is of great importance since 5-10% of infected adults will not clear the infection after the initial phase of the illness. About 25% of people who do not initially clear the infection will later develop chronic active hepatitis.

This study will evaluate the safety and immunogenicity of HEPLISAV™ when administered to adults who have end-stage renal disease (glomerular filtration rate [GFR] ≤ 45 mL/min). Once subjects have been consented, screened, and randomized to treatment, subjects will receive a total of three injections over a 24-week period, with follow-up visits at 28 and 50 weeks. Subjects will receive 1 of the following 2 regimens:

* HEPLISAV™ single dose at Day 0, 4 weeks (1 month) and 24 weeks (6 months)
* HEPLISAV™ double dose at Day 0, 4 weeks (1 month) and 24 weeks (6 months)

Safety and tolerability will be evaluated by occurrence of adverse events, periodic laboratory tests, vital signs, and local and systemic reactogenicity.

Immunogenicity will be evaluated by the proportion of subjects exhibiting a seroprotective immune response (anti-hepatitis B surface antigen antibodies [anti-HBsAg] ≥ 10 milli-international unit (mIU)/mL) at Weeks 4, 12, 24, 28 and 50.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent
* Have a glomerular filtration rate (GFR) ≤ 45 mL/min
* Have an expectation of going on hemodialysis or are already on hemodialysis
* Is serum negative for hepatitis B virus (HBV) antibodies, hepatitis C virus (HCV), and human immunodeficiency virus (HIV)
* Have repeated resting blood pressure measurements ≤ 165/105 mmHg
* Women of childbearing potential must be consistently using a highly effective method of birth control

Exclusion Criteria:

* Women who are pregnant, breastfeeding or planning a pregnancy
* Any previous HBV infection
* Previous vaccination (1 or more doses) with any HBV vaccine
* Any previous autoimmune diseases
* Have a diagnosis of chronic renal failure due to autoimmune disease
* Are at high risk for recent exposure to HBV, HCV or HIV
* Received any antibodies within 3 months prior to study entry
* Ever received an injection with DNA plasmids or oligonucleotides
* Received any vaccines within 4 weeks prior to study entry
* Received any other investigational medicinal agent within 4 weeks prior to study entry

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-07; Primary Completion 2008-08 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events and local and systemic reaction rates | 28 weeks

SECONDARY OUTCOMES:
Portion of subjects who have a seroprotective immune response (anti-HBsAg ≥ 10 mIU/ml) | 50 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Martins, MD, D Phil, Study Director — Dynavax Technologies Corporation
Locations (3):
- Canada (3):
  - White Hills Medical Clinic, St. John's, Newfoundland and Labrador
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - SMBD - Jewish General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Dynavax Webpage — http://www.dynavax.com